CLINICAL TRIAL: NCT04646551
Title: Assessment of the Pattern and Risk Factors of Covid-19 Between Infected Healthcare Workers at Assiut University Hospitals
Brief Title: Covid-19 Risk Factors and Pattern Between Healthcare Workers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sahar Ahmed, Sahar Ahmed okily Ahmed, Assiut University
Other Study IDs: Covid-19 patterrn
Record Dates: First submitted 2020-11-26; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Assessment of the Pattern and Risk Factors of Covid-19 between infected Healthcare Workers at Assiut University Hospitals

DETAILED DESCRIPTION:
COVID-19 is a respiratory infectious disease caused by a novel coronavirus, SARS-CoV-2. The first batch of COVID-19 patients were found in December 2019 (1). The disease is mainly transmitted through respiratory droplets and close contact, and all people are susceptible to it (2). SARS-CoV-2 is highly contagious (3), and has quickly spread to most countries and regions of the world. COVID-19 has become a global pandemic and has received great attention from all over the world (4, 5). Till April 7, 2020, 1,214,466 confirmed cases of COVID-19 have been found in 211 countries and regions, causing 67,767 deaths (6). The main clinical manifestations of COVID-19 are cough, fever, malaise, chest distress and tachypnia and complications such acute respiratory distress syndrome.

Healthcare workers (HCWs) are on front line of treating patients infected with COVID-19. However, data related to infection rate among HCWs are limited. Early available evidence suggested that HCWs are being increasingly infected with the novel infection ranging from 15% to 18% and in some cases up to 20% of the infected population. Major risk factors of infection among HCWs include lack of understanding of the disease, inadequate use and availability personal Protective Equipment (PPE), uncertain diagnostic criteria, unavailability of diagnostic tests and psychological stress. Therefore the protection of HCWs by authorities should be prioritized through education and training, the readiness of staff, incentives, availability of PPEs, and psychological support. In this time of COVID-19 pandemic, big problem in hospitals that are flooded with infected symptomatic and asymptomatic patients. A critical aspect is the protection of the HCWs who are at risk, including individuals more than 50 years old those with presence of a systemic disease, smokers and disabled individuals. These HCWs should be identified and not assigned duties inwards and premises managing COVID 19 patients

ELIGIBILITY:
Inclusion Criteria:

- Health care workers in Assiut University Hospitals ( ≥ 18 years old) who were infected with covid-19 and were diagnosed based on either PCR testing or based on radiological diagnosis.

Those who were not in contact with household Covid-19 patients within 14 days before getting infected.

Those who were adherent to social isolation apart from their work

b. Exclusion criteria : Patients with Covid-19 who are not HCWs in Assiut University Hospital. Those who were in contact with household infected patients within 14 days before getting infected.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthcare Workers
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the Pattern and Risk Factors of Covid-19 between infected Healthcare Workers | Baseline
  Risk Factors of Covid-19

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mostafa Abdelhady, Study Director — Professor

IPD SHARING:
Plan to Share IPD: No